CLINICAL TRIAL: NCT00215072
Title: Death Following Congenital Heart Surgery
Status: Terminated | Type: Observational
Why Stopped: insufficient number of patient charts to support hypothesis
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-090
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Heart Surgery; Congenital Heart Defects
Keywords: Death after heart surgery; surgical mortality; post-operative mortality; pediatric health; cardiac
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to elucidate the patterns of death following congenital heart surgery.

DETAILED DESCRIPTION:
With the improvements in instrumentation, surgical technique, and critical care, the overall mortality following congenital heart surgery has become extremely low. Also, with the introduction of extracorporeal support (ECMO), especially in the emergency setting, acute deaths are extremely rare. The majority of post-operative deaths seem to be the result of a prolonged hospitalization with a progressive decline to multi-system organ failure.

The primary aim of the study is to elucidate the patterns of death following congenital heart surgery. The secondary aims of the study are to discover patterns and consistencies among the deaths and to discover points of potential intervention to reduce surgical mortality. The study will be conducted through a retrospective chart review of approximately 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the congenital surgery database
* Post-operative surgical mortality
* Deaths within 30 days of surgery
* Deaths prior to ever leaving the hospital

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in the congenital surgery database
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2005-07; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States